CLINICAL TRIAL: NCT01973790
Title: A Phase III, Multicentre, Single-arm, Open-label Study to Evaluate the Long-term Safety of Z-338 in Subjects With Functional Dyspepsia
Brief Title: Phase III, Long-term, Open-label Safety Study of Z-338
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z338-01
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-01

CONDITIONS: Dyspepsia
Keywords: Z-338; Functional Dyspepsia; Postprandial Distress Syndrome
MeSH Terms: conditions — Dyspepsia | interventions — Z 338

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Z-338 (Experimental): 100mg TID
  Interventions: Drug: Z-338

INTERVENTIONS:
Drug: Z-338 — 100mg TID
  Other Names: Acotiamide

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of 100 mg Z-338 TID in European subjects with FD.

DETAILED DESCRIPTION:
This is a Phase III, multicentre, single-arm, open-label study to evaluate the long-term safety of 100 mg Z-338 TID in subjects with FD.

The study comprises a screening period (up to 3 weeks), a run-in period (1 week) and an open-label treatment period (52 weeks). Including an additional 2-week follow-up period for assessment of AEs, the maximum duration of a subject's participation in the study will be 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to provide written informed consent prior to any study procedures being performed
* Subjects with a diagnosis of FD (postprandial distress syndrome) as defined by the Rome III Criteria
* Subjects must present Postprandial Fullness or Early Satiation as the most bothersome symptom during the 6 months prior to informed consent.
* Subjects must have a normal endoscopy result within the 6 months (3 months in case of subjects who are Helicobacter pylori positive) prior to informed consent or during the screening period.

Exclusion Criteria:

* Subjects on PPI(s) who are unable to discontinue PPI medication by the end of the screening period
* Subjects taking drugs that affect gut motility, gut sensitivity and/or acid secretion who are unable to discontinue these drugs by the end of the screening period
* Subjects who have received H. pylori eradication therapy during the 3 months prior to informed consent
* Subjects with confirmed organic gastrointestinal disease
* Subjects presenting with predominant complaints relieved by stool movements (irritable bowel syndrome)
* Subjects presenting with predominant GORD symptoms
* Subjects presenting with predominant complaints of chronic idiopathic nausea
* Subjects with Type I or Type II diabetes
* Subjects with body mass index (BMI) over 30 kg/m2
* Subjects with any condition which, in the opinion of the Investigator, makes the subject unsuitable for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
General safety endpoints | up to 58 weeks
  Adverse Events, 12-lead ECGs, Laboratory variables, Vital signs, Physical examination

SECONDARY OUTCOMES:
To explore the efficacy | up to 52 weeks
  the use of LPDS to measure FD symptom severity and the effect of Z-338, the effect of Z-338 on the QoL in subjects with FD as measured by SF-36 survey and SF-NDI, the effect of Z-338 on work productivity in subjects with FD as measured by WPAI.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — University of Leuven, University Hospital Gasthuisberg
Locations (36):
- Zeria Investigative site, Leuven, Belgium
- Bulgaria (3):
  - Zeria Investigative Site, Plovdiv
  - Zeria Investigative Sites, Sofia
  - Zeria Investigative site, Varna
- Latvia (3):
  - Zeria Invetigative Site, Liepāja
  - Zeria Investivgative SIte, Limbaži
  - Zeria Investigative Sites, Riga
- Lithuania (4):
  - Zeria Investigative Site, Alytus
  - Zeria Investigative Sites, Kaunas
  - Zeria Investigative Site, Klaipėda
  - Zeria Investigative Site, Vilnius
- Romania (6):
  - Zeria Investigative Site, Brasov
  - Zeria Investigative Sites, Bucharest
  - Zeria Investigative Sites, Cluj-Napoca
  - Zeria Investigative Site, Sibiu
  - Zeria Investigative Site, Târgu Mureş
  - Zeria Investigative Sites, Timișoara
- Russia (4):
  - Zeria Investigative Site, Kazan'
  - Zeria Investigative Site, Ryazan
  - Zeria Investigative Site, Saratov
  - Zeria Investigative Site, Yaroslavl
- Slovakia (7):
  - Zeria Investigative sites, Bratislava
  - Zeria Investigative sites, Košice
  - Zeria Investigative Site, Malacky
  - Zeria Investigative Site, Martin
  - Zeria Investigative Site, Nitra
  - Zeria Investigative Site, Prešov
  - Zeria Investigative Site, Trnava
- Sweden (2):
  - Zeria Investigative Site, Gothenburg
  - Zeria Investigative Sites, Stockholm
- Ukraine (3):
  - Zeria Investigative Site, Dnipropetrovsk
  - Zeria Investigative Site, Kyiv
  - Zeria Investigative Site, Vinnytsia
- United Kingdom (3):
  - Zeria Investigative site, Barnstaple
  - Zeria Investigative site, Bath
  - Zeria Investigative Site, Royal Leamington Spa

REFERENCES:
- [Derived] Tack J, Pokrotnieks J, Urbonas G, Banciu C, Yakusevich V, Bunganic I, Tornblom H, Kleban Y, Eavis P, Tsuchikawa M, Miyagawa T. Long-term safety and efficacy of acotiamide in functional dyspepsia (postprandial distress syndrome)-results from the European phase 3 open-label safety trial. Neurogastroenterol Motil. 2018 Jun;30(6):e13284. doi: 10.1111/nmo.13284. Epub 2018 Jan 8. PMID 29315999